CLINICAL TRIAL: NCT00691535
Title: Association of BDNF, COMT, MDRI, CRH, CRF, and GC Receptor Genetic Polymorphisms With Symptomatology and Treatment Response in Psychotic Major Depression
Brief Title: Genetics of Symptomatology and Treatment Response in Psychotic Major Depression
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alan Schatzberg, Principle Investigator, Stanford University
Other Study IDs: SU-05132008-1160
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Psychotic Disorders; Depressive Disorder; Depressive Disorder, Major
MeSH Terms: conditions — Psychotic Disorders; Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
We hope to learn more about the biology of psychiatric illness with the hope of improving the diagnosis and treatment of such psychiatric conditions as major depression.

DETAILED DESCRIPTION:
From the blood sample you donate, the researchers will obtain DNA. This DNA will be used to search for DNA markers related to the underlying biology of psychiatric illness and how this might explain the symptoms of these disorders. Research using DNA is an important way to try to understand human disease and/or the role genes play in disease. In effect, part of your blood sample will be used to attempt to understand how genetic factors contribute to the symptoms of such psychiatric conditions as major depression.

ELIGIBILITY:
Inclusion Criteria:

1. You are currently experiencing symptoms that are consistent with an episode of major depression without symptoms of psychosis (such as hallucinations, delusions or disorder of thought process), or
2. You are currently experiencing symptoms that are consistent with an episode of major depression with symptoms of psychosis (such as hallucinations, delusions or disorder of thought process), or
3. You have been diagnosed with either schizophrenia or schizoaffective disorder, or
4. You are a volunteer without a history of psychiatric illness (a healthy control subject).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 2003-10 (Actual); Primary Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan F Schatzberg, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States